CLINICAL TRIAL: NCT06857175
Title: A Phase III Randomized Controlled Clinical Study Comparing BL-B01D1 With Chemotherapy of Physician's Choice in Patients With Recurrent or Metastatic Urothelial Carcinoma After Failure of PD-1/PD-L1 Monoclonal Antibody and Platinum-based Chemotherapy
Brief Title: A Study Comparing BL-B01D1 With Chemotherapy of Physician's Choice in Patients With Recurrent or Metastatic Urothelial Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-309
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Docetaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-B01D1 (Experimental): Participants receive BL-B01D1 in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1
- Docetaxel or Paclitaxel (Active Comparator): Participants receive Docetaxel or Paclitaxel in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Docetaxel or Paclitaxel

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
  Arms: BL-B01D1
Drug: Docetaxel or Paclitaxel — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Docetaxel or Paclitaxel

SUMMARY:
This trial is a registered phase III, randomized, open-label and multicenter study to evaluate the efficacy and safety of BL-B01D1 in patients with recurrent or metastatic urothelial carcinoma after failure of PD-1/PD-L1 monoclonal antibody and platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Age: ≥18 years old;
3. Expected survival time ≥3 months;
4. Patients with unresectable locally advanced or metastatic urothelial carcinoma who had failed platinum-based chemotherapy and PD-1/PD-L1 inhibitors;
5. Patients with locally advanced or metastatic urothelial carcinoma who are eligible for treatment with the control chemotherapy agents specified in this protocol;
6. Consent to provide archival tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 3 years;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. ECOG 0 or 1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. If blood transfusion and colony-stimulating factor were not allowed within 14 days before randomization, the organ function level had to meet the requirements;
12. A serum pregnancy test must be performed within 7 days before the start of treatment for premenopausal women of childbearing potential, and the result must be negative and must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Chemotherapy, targeted therapy, biological therapy, etc. were used within 4 weeks or 5 half-lives before randomization;
2. Patients with locally advanced or metastatic urothelial carcinoma who were suitable for radical local therapy were excluded;
3. Frontline received ADCs targeting topoisomerase I inhibitors or EGFR and/or HER3; The front line had received both paclitaxel and docetaxel;
4. History of severe heart disease and cerebrovascular disease;
5. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis was excluded;
6. Prolonged QT interval, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
7. Diagnosed with active malignancy within 3 years before randomization;
8. Hypertension poorly controlled by two antihypertensive drugs (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
9. Patients with poor glycemic control;
10. Patients with grade ≥1 radiation pneumonitis according to the RTOG/EORTC definition; Previous history of ILD, or suspicion of such disease during screening;
11. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
12. Patients with active central nervous system metastases;
13. Severe infection occurred within 4 weeks before randomization; Evidence of pulmonary infection or active pulmonary inflammation within 2 weeks before randomization;
14. Patients with massive or symptomatic effusions or poorly controlled effusions;
15. Imaging examination indicated that the tumor had invaded or wrapped around the large blood vessels of the abdomen, chest, neck, and pharynx, except for those that the investigator thought would not affect the patient's enrollment in the drug;
16. Serious unhealed wound, ulcer or fracture within 4 weeks before signing the informed consent;
17. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
18. Patients with inflammatory bowel disease, extensive bowel resection, immune enteritis, intestinal obstruction or chronic diarrhea;
19. Patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of BL-B01D1;
20. Had a history of autologous or allogeneic stem cell transplantation;
21. Human immunodeficiency virus antibody positive, active hepatitis B virus infection or hepatitis C virus infection;
22. A history of severe neurological or psychiatric illness;
23. Received other unmarketed investigational drugs or treatments within 4 weeks before randomization;
24. Subjects who were scheduled to be vaccinated or received live vaccine within 28 days before study randomization;
25. Other circumstances in which the investigator considered it inappropriate to participate in the trial because of complications or other circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China